CLINICAL TRIAL: NCT06961526
Title: Primary Prophylaxis of Esophageal Varices in Patients Treated With Atezolizumab and Bevacizumab for Advanced Hepatocellular Carcinoma.
Brief Title: Esophageal Varices Prophylaxis in Hepatocellular Carcinoma Treated With Atezolizumab and Bevacizumab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36264PR1125/3/25
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Esophageal and/or Gastric Varices; Hepatocellular Carcinoma (HCC)
Keywords: Esophageal varices; hepatocellular carcinoma; atezolizumab-bevacizumab therapy
MeSH Terms: conditions — Esophageal and Gastric Varices; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCC patients with small non-risky EGVs (Active Comparator): 55 patients with small EGVs that had no red signs undergoing variceal band ligation.
  Interventions: Procedure: Esophageal band ligation
- HCC patients with no or small non-risky EGVs (No Intervention): 55 patients with no or small EGVs that had no red signs. patients will be followed up after 3, 6, 9, 12 months of atezolizumab-bevacizumab therapy.

INTERVENTIONS:
Procedure: Esophageal band ligation — upper endoscopy will be performed within 6 months before starting atezolizumab-bevacizumab therapy in HCC patients. Esophageal band ligation for small non-risky varices before starting atezolizumab-bevacizumab therapy. Endoscopy will be repeated 3, 5, 9, 12 months after atezolizumab-bevacizumab therapy
  Arms: HCC patients with small non-risky EGVs

SUMMARY:
The goal of this prospective cohort study is to evaluate the progression of esophagogastric varices in patients treated with atezolizumab-bevacizumab. Assess the efficacy of primary prophylaxis of small esophageal varices with no risky signs and shortening endoscopic follow-up time intervals to reduce the risk of variceal hemorrhage.

Researchers will assess the progression of esophageal varices (EVs) with no bleeding stigmata in patients treated with atezolizumab-bevacizumab therapy at 3, 6, 9, and 12 months with endoscopic examination. Evaluate the effect of shortening the endoscopic follow-up intervals to reduce the risk of variceal bleeding in patients treated with atezolizumab-bevacizumab therapy. Researchers will also assess the efficacy of variceal band ligation in small varices without bleeding stigmata before starting atezolizumab-bevacizumab therapy to reduce the progression of EVs.

Participants will undergo history-taking, clinical examination, laboratory investigations, Triphasic CT abdomen with contrast or MRI (for evaluation of tumor site, size and number), abdominal ultrasonography, and upper endoscopy (within 6 months before beginning of systemic therapy and followed up after 3, 6, 9, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed advanced HCC (Diagnosed by two imaging modalities or liver biopsy) eligible for atezolizumab-bevacizumab therapy.
* Patients with preserved liver function (compensated Child-Pugh A if there is underlying cirrhosis).
* Patients with performance status ≤2 at staging work-up.
* Patients with no or grade 1 non-risky esophageal varices on pretreatment endoscopic examination.

Exclusion Criteria:

* Child-Pugh class C patients.
* Patients with performance status >2 at staging work-up.
* Vascular disorders and arterial hypertension.
* Severe autoimmune disorders.
* Patients who lost follow-up.
* Pregnant or breastfeeding women.
* Unwilling to participate in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
esophagogastric varices progression rate | through study completion, an average of 1 year
  evaluating esophagogastric varices progression rate at 3, 5, 9, and 12 months of starting atezolizumab-bevacizumab therapy.
variceal band ligation in small varices without bleeding stigmata | through study completion, an average of 1 year
  Evaluating the effect of variceal band ligation in small varices without bleeding stigmata in reducing the variceal bleeding rate.

SECONDARY OUTCOMES:
shortening the endoscopic follow-up intervals | through study completion, an average of 1 year
  Evaluating the effect of shortening the endoscopic follow-up intervals to reduce the variceal bleeding rate in patients treated with atezolizumab-bevacizumab therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Elkafoury, MD, Principal Investigator — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt